CLINICAL TRIAL: NCT04654728
Title: Prospective Randomized Study Comparing ePTFE Versus Dacron Graft Donor Liver Transplantation
Brief Title: Prospective Randomized Study Comparing ePTFE Versus Dacron Graft for Anterior Sector Venous Drainage in Right Lobe Living Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ATIF TEKIN, General Surgery Residence, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medipol Transplant
Record Dates: First submitted 2020-11-23; First posted 2020-12-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Patency and Infection Rates Due to Usage of PTFE vs.Dacron Grafts

STUDY DESIGN:
Intervention Model Description: Patients will be equally randomized into two groups using sealed envelope system. For anterior sector venous drainage, ePTFE vascular grafts (straight or bifurcated) in group 1, and Dacron grafts(straight or bifurcated) in 2 will be used as conduit.
Masking Description: None(Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ePTFE graft (Active Comparator): In this group, anterior sector of the right lobe graft will be reconstructed using ePTFE vascular grafts
  Interventions: Procedure: Active Comparator: ePTFE graft
- Dacron graft (Other): In this group, anterior sector of the right lobe graft will be reconstructed using Dacron vascular grafts
  Interventions: Procedure: Active Comparator: ePTFE graft

INTERVENTIONS:
Procedure: Active Comparator: ePTFE graft — In this group, anterior sector of the right lobe graft will be reconstructed using Dacron vascular grafts
  Other Names: Other: Dacron graft

SUMMARY:
Living donor liver transplantation (LDLT) using the right lobe (RL) has created a significant increase in graft supply worldwide. However, it is a technically demanding procedure particularly because of the unique functional anatomic characteristics of hepatic venous drainage [1].

DETAILED DESCRIPTION:
In the absence of an adequate drainage of the anterior sector (AS) veins, the consequent venous congestion in the RL graft may result in impaired graft regeneration, immediate liver dysfunction, and graft loss even in a liver graft of adequate size [2]. To overcome this problem, Lee et al. [3] introduced the concept of modified RL graft in which the branches of the middle hepatic vein (MHV) was drained using interposition vascular grafts. Although, the issue of when and how the MHV branches should be drained has been controversial since then, reconstruction of segment 5 and 8 veins using an interposition graft has become a standard procedure during RL LDLT. The vascular graft of choice in this procedure has been cryopreserved homologous vein graft, which provides excellent patency with low infection risk. However, such grafts are often unavailable, particularly in programs where deceased donors are scarce and surgeons must rely on synthetic grafts such as expanded polytetrafluoroethylene (ePTFE) and polyethylene terephthalate (Dacron®). Since we have developed an "intent-to-drain" policy in our LDLT program, we have been using Dacron grafts exclusively [4]. Although, complications such as early graft thrombosis, graft infection, and hollow viscous migration remain as major concerns, the safety and efficacy of both ePTFE and Dacron grafts in LDLT has been proven [5, 6]. However, to date, none of the previous studies have specifically compared these two different prosthetic materials, addressing graft patency and complication rates in patients undergoing LDLT. The aim of our study is to compare AS venous outflow reconstruction using ePTFE vs. Dacron grafts for their patency and infection rates and outcomes with respect to graft and patient survival in RL LDLT.

ELIGIBILITY:
Inclusion Criteria:

1. Primary Adult Living Donor Liver Transplantation
2. Right Lobe graft with anterior sector venous outflow reconstruction -

Exclusion Criteria:

1. Right Lobe graft without anterior sector venous outflow reconstruction
2. Liver re-transplantation -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Graft patency at 6-month posttransplant | 6 months
  Graft Patency

SECONDARY OUTCOMES:
Graft-related complications | One Year
  Rate of graft infection
Graft survival | One year
  Morbidity
Patient survival | One Year
  Mortality
Graft regeneration rate | 6 months
  Graft regeneration

CONTACTS AND LOCATIONS:
Overall Officials: Murat Dayangac, M.D., Study Director — Study Chief
Locations (1):
- Medipol University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No